CLINICAL TRIAL: NCT00483210
Title: Tissue Lipids and Insulin Resistance
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The study goals were accomplished by a similar study at UAMS. (W.J. Evans)
Sponsor: University of Arkansas (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Carole Hamon, University of Arkansas for Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 72495
Record Dates: First submitted 2007-06-04; First posted 2007-06-06 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2015-03

CONDITIONS: Tissue Lipid Metabolism
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Fenofibrate

SUMMARY:
Resistance to the hypoglycemic action of insulin develops within 7 days of bedrest in young, healthy volunteers. We propose that the same event occurs in elderly individuals confined to bed, that alterations in lipid metabolism are, at least in part, responsible for the insulin resistance associated with bedrest, and that the accumulation of intracellular triglyceride (TG) in liver and muscle will play a role in impairing insulin action. Further, we propose that the PPARα (Peroxisome Proliferator-Activated Receptor Alpha) agonist fenofibrate will increase tissue fatty acid disposal by activating mitochondrial oxidative capacity, thereby improving insulin sensitivity.

We will investigate a series of specific hypotheses designed to examine the role of altered lipid metabolism in the development of insulin-resistance associated with bedrest. Further, since inactivity is likely a principal factor in the development of insulin resistance in the elderly, the response to the inactivity imposed by bedrest represents an acceleration of the normal development of insulin resistance in elderly individuals. Therefore, the results of this study will also be pertinent to the understanding of the mechanisms responsible for the natural development of insulin resistance in free-living elderly.

DETAILED DESCRIPTION:
The accumulation of intracellular lipid reflects a dysregulation of tissue fatty acid metabolism involving abnormal relationships between tissue fatty acid uptake and oxidation. It has been postulated that such dysregulation of lipid metabolism causes insulin resistance as a direct consequence of the accumulated intracellular triglyceride (TG), or that the increased intracellular TG reflects an increase in active products of fatty acids, such as diacylglycerol, that inhibit the insulin signaling pathway. We recently found that both muscle and liver intracellular TG concentrations were elevated in more than one-half of otherwise healthy elderly individuals.

We hypothesize that an increase in tissue lipids in the elderly reflects altered tissue lipid metabolism that puts them at high risk for the development of insulin resistance with bedrest. Further, we propose that the PPARα (Peroxisome Proliferator-Activated Receptor Alpha) agonist fenofibrate will increase tissue fatty acid disposal by activating mitochondrial oxidative capacity, thereby improving insulin sensitivity.

We will examine the role of alterations in lipid metabolism in the development of insulin resistance that occurs with bedrest.

Methods: A total of 40 elderly subjects ranging in age from 60-85 will be studied. Subjects will be randomized to one of two groups: 1) 10 days of bedrest or 2) 10 days of bedrest plus fenofibrate. Each of the subjects will complete a 5- day diet stabilization period and have a metabolic infusion study on day 5, followed by 10 days of bedrest and a metabolic study on day 18. This will be followed by a 3 week rehabilitation program. Pre-test and post bedrest measurements include body composition by DEXA, intracellular TG measurements by MRS, strength testing.

The results will provide insight into the mechanisms responsible for the development of insulin resistance with inactivity and strategies for ameliorating this response.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 60 and 85
* Availability of transportation
* Ability to sign informed consent and a score >24 on the 30-item Mini-Mental Status Exam

Exclusion Criteria:

* Subjects with limiting or unstable angina or a cardiology confirmed ECG which demonstrates cardiac abnormalities such as >0.2mV horizontal or downsloping ST segment depression, frequent arrhythmia's (>10PVC/min), or valvular disease.
* Subjects with vascular disease as determined by a combination of risk factors of peripheral atherosclerosis, uncontrolled hypertension, obesity, uncontrolled diabetes, or hypercholesterolemia >250mg/dl.
* Any subjects taking Coumadin adn risk factors of DVT as listed:

  1. previous incidents of diagnostically verified DVT
  2. major orthopedic, thoracic, abdominal, genitourinary surgery within the last 6 months
  3. traumatic fractures of pelvis, femur, or tibia
  4. prolonged immobilization: paralysis, pareses or plaster immobilization of lower extremities or prolonged bed rest within the last 6 months
  5. estrogen use: estrogen substitution/supplementation within the last 6 months
  6. venulitis, thromboangitis obliterans, homocyteinuria within the last 3 months
  7. known hypercoagulative abnormalities
  8. more than 1 point on the DVT risk assessment score
* Subjects with low hemoglobin or hematocrit (i.e., lower than accepted lab values)
* Any subject that has a chronically elevated systolic pressure >170 or a diastolic pressure >100 will be excluded. Subjects may be included if they are taking blood pressure medication and have a blood pressure below these criteria.
* Any subject that is HIV-seropositive, or has active hepatitis.
* Any subject with an uncontrolled metabolic disease including liver or renal disease.
* Any subject currently taking aspirin that cannot be discontinued for medical reasons.
* Presence of acute illness or metabolically unstable chronic illness.
* Any subject currently on weight-loss diet.
* Inability to abstain from smoking for duration of study.
* Recent ingestion of anabolic steroids or corticosteroids(within 3 months)
* Subjects with atrial fibrillation, history of syncope, angina, or congestive heart failure.
* Subjects with cancer or recently (6 months) treated cancer other than basal cell carcinoma.
* Body mass index greater than 35 or less than 20kg/m2.
* Score of less than 9 on Guralnik/EPESE Scale.
* Any known hypersensitivity to or allergy to fenofibrate.
* Any other condition or event considered exclusionary by the PI and covering faculty physician.

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wolfe, PhD, Principal Investigator — University of Arkansas